CLINICAL TRIAL: NCT04041518
Title: Autotransplantation of Teeth With Advanced or Completed Root Development With Intraoperative Extra-corporal Apicoectomy
Brief Title: Autotransplantation of Teeth With Intraoperative Extra-corporal Apicoectomy
Acronym: ZahnTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30-519 ex 17/18
Record Dates: First submitted 2019-07-17; First posted 2019-08-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Missing Tooth
Keywords: Autotransplantation; extraoral apicoectomy; revascularization
MeSH Terms: conditions — Anodontia | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Autotransplantation and intra-operative extraoral apicoectomy of a permanent tooth.
  Interventions: Procedure: Autotransplantation

INTERVENTIONS:
Procedure: Autotransplantation — Autotransplantation of tooth with an almost fully or completely developed root with intraoperative extraoral apicoectomy.

SUMMARY:
Clinical trial to evaluate the success rate of autotransplantation of teeth with advanced or completed root growth with intraoperative extracorporeal root tip resection in 20 patients.

DETAILED DESCRIPTION:
Autotransplantation is surgical transposition of a tooth by extraction and replantation into another site in the same patient's mouth. It has become a routine treatment option for missing teeth in the human dentition and a reasonable alternative to dental implants, fixed bridgework, resin-bonded restorations, and removable partial dentures.

Under ideal circumstances, a vital transplanted tooth with healthy periodontal tissues is the final outcome of autotransplantation. Best results for both the rate of revascularization and the further development of the roots are achieved in adolescent teeth with two thirds to three fourths developed roots. According to Andreasen et al., the critical diameter of the apical foramen of the transplanted tooth is 1 mm for successful revascularization. The reported success rates for revascularization of mature teeth with fully developed roots were distinctly lower, and endodontic treatment was considered a standard procedure after transplantations of mature teeth.

Aim of the presented study is to evaluate the success rate of autotransplantation of almost or completely fully developed teeth with intraoperative extracorporeal root tip resection to facilitate revascularization and obviate subsequent root canal treatment.

The primary endpoint is the successful periodontal healing of the graft, the secondary endpoint the revascularization of the graft.

Revascularization is assessed radiologically with intraoral films after four weeks and three, six, nine and twelve months (obliteration of the pulp, no signs of inflammatory root resorption, and magnetic resonance tomography 4 weeks postoperatively.

Patients are followed-up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Male and female consenting and judicious young people and adults
* Written consent of the participant and, if applicable, of the legal guardian after education
* Planned tooth transplantation with advanced or completed root growth

Exclusion Criteria:

Contrast agent allergy (Gadovist®)

* Contraindications for magnetic resonance imaging (MRI): (pronounced metal restorations, running orthodontics with metal, fixed appliance in the target jaw)
* Current or past antiresorptive therapy with bisphosphonates
* Further anamnestic general or local risk situation, among others:

Anti-angiogenic therapy, History of local radiation therapy, severe coagulation disorder, unadjusted diabetes mellitus, malignant diseases

* Acute gingivitis or advanced periodontitis
* Participation in an ongoing drug trial (various drugs may distort the result, such as bisphosphonates, cortisone, chemotherapeutics, angiogenesis inhibitors)
* heavy smokers (> 10 per day)
* Acute or chronic infections (osteomyelitis) at the surgical site
* metabolic diseases (diabetes, hyperparathyroidism, osteomalacia)
* Severe kidney dysfunction, severe liver disease
* Patients with high-dose corticosteroid therapy
* prolonged corticosteroid or radiotherapy in the oral cavity
* autoimmune diseases
* Pregnant or breastfeeding women

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Periodontal Healing | 3 to 12 months
  Formation of a healthy periodontal ligament with no signs of ankylosis and normal tooth mobility, assessed with electromechanical tapping and intraoral radiography

SECONDARY OUTCOMES:
Revascularization | 2 months
  Restoration of the circulation of the pulp, assessed with Magnetic resonance imaging and intraoral radiography
Re-innervation | 3, 6, 9 and 12 months
  Restoration of Sensitivity of the pulp, assessed with electric pulp testing

CONTACTS AND LOCATIONS:
Overall Officials: Petra Rugani, DDS, Principal Investigator — Medical University of Graz; Petra Rugani, DDS, Study Director — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakse N, Ruckenstuhl M, Rugani P, Kirnbauer B, Sokolowski A, Ebeleseder K. Influence of Extraoral Apicoectomy on Revascularization of an Autotransplanted Tooth: A Case Report. J Endod. 2018 Aug;44(8):1298-1302. doi: 10.1016/j.joen.2018.04.016. Epub 2018 Jun 20. PMID 29935869